CLINICAL TRIAL: NCT05069207
Title: EVALUATION OF DIAPRAGMATIC BREATHING IN POSTURAL STABILIZATION IN CHILDREN WITH URINARY INCONTINENCE
Brief Title: The Effect of the Diaphragm in Urinary Incontinence
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Sümeyra Kapucu, physiotherapist, Kırıkkale University
Other Study IDs: KırıkkaleUniversity71
Record Dates: First submitted 2021-09-16; First posted 2021-10-06 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-03

CONDITIONS: Urinary Incontinence
Keywords: diaphragmatic breathing
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Monosymptomatic Enuresis: Quality of Life Scale in Children with Urinary Incontinence (PIN-Q) Voiding Disorders Symptom Score (IBSS) Dynamic Neuromuscular Stabilization (DNS) Maximum inspiratory pressure (MIP) and volume (Volume (V)) parameters will be evaluated with the POWER breathe K5 to evaluate
  Interventions: Other: POWER breathe K5
- Non-monosymptomatic Enuresis: Quality of Life Scale in Children with Urinary Incontinence (PIN-Q) Voiding Disorders Symptom Score (IBSS) Dynamic Neuromuscular Stabilization (DNS) Maximum inspiratory pressure (MIP) and volume (Volume (V)) parameters will be evaluated with the POWER breathe K5 to evaluate
  Interventions: Other: POWER breathe K5
- Daytime Urinary Incontinence: Quality of Life Scale in Children with Urinary Incontinence (PIN-Q) Voiding Disorders Symptom Score (IBSS) Dynamic Neuromuscular Stabilization (DNS) Maximum inspiratory pressure (MIP) and volume (Volume (V)) parameters will be evaluated with the POWER breathe K5 to evaluate
  Interventions: Other: POWER breathe K5
- Control Group Healthy Individuals: Quality of Life Scale in Children with Urinary Incontinence (PIN-Q) Voiding Disorders Symptom Score (IBSS) Dynamic Neuromuscular Stabilization (DNS) Maximum inspiratory pressure (MIP) and volume (Volume (V)) parameters will be evaluated with the POWER breathe K5 to evaluate
  Interventions: Other: POWER breathe K5

INTERVENTIONS:
Other: POWER breathe K5 — Maximum inspiratory pressure (MIP) and volume (Volume (V)) parameters will be evaluated with the POWER breathe K5 to evaluate

SUMMARY:
Urinary incontinence in children is defined as involuntary leakage of urine. Urinary incontinence is the most common urological complaint in children. Many factors are effective in urinary incontinence. Research on the effectiveness of the diaphragm in postural stabilization, which the investigators think is one of these factors, is limited. The aim of this study is to compare the effectiveness of diaphragmatic breathing in postural stabilization with healthy individuals and individuals with urinary incontinence. As a result, it has been revealed that one factor of urinary incontinence is due to the dysfunction of diaphragmatic breathing and will be a step to increase awareness on diaphragmatic breathing.

DETAILED DESCRIPTION:
Urinary incontinence in children is defined as involuntary leakage of urine. Urinary incontinence is the most common urological complaint in children. Nocturnal incontinence is the most common chronic problem of childhood as well as allergic diseases. Frequency rates of 5-15% are reported in various sources, and in studies conducted with school children in our country, quite high rates of 20-30% are found. It is estimated that there are over 50 million children with urinary incontinence worldwide.

There are many studies in the literature to determine the epidemiology and causes of urinary incontinence. In this study, it is aimed to evaluate diaphragmatic breathing in postural stabilization in children with urinary incontinence. In our study, Kırıkkale University Faculty of Medicine hospital; Individuals between the ages of 5 and 18 who were diagnosed with urinary incontinence and volunteered to participate in the study will be included in the study. The number of individuals will be determined according to the power analysis to be made. Individuals will be divided into 4 groups according to their diagnosis. Four groups with monosymptomatic enuresis, non-monosymptomatic enuresis, daytime urinary incontinence and healthy children as the control group will be included in the study. Before individuals; Demographic characteristics such as age, gender, height and weight will be questioned.

Quality of Life in Children with Urinary Incontinence Scale (PIN-Q), which is the evaluation parameters of the children included in the study, Voiding Disorders Symptom Score (IBSS) to assess the severity of children's voiding disorder symptoms , Dynamic Neuromuscular stabilization (DNS) to evaluate the diaphragm in postural stabilization ; S-index (Inspiratory muscle strength), Maximum inspiratory pressure (MIP) and volume (Volume (V)) parameters will be evaluated with the POWER breathe K5 to evaluate.

Hypotheses :

H01: Diaphragmatic breathing is active in postural stabilization in children with monosymptomatic enuresis compared to healthy children.

H02: Diaphragmatic respiration is active in postural stabilization in children with non-monosymptomatic enuresis compared to healthy children.

H03: Diaphragmatic breathing is active in postural stabilization in children with daytime urinary incontinence compared to healthy children.

H1: In children with monosymptomatic enuresis, diaphragmatic breathing is not active in postural stabilization compared to healthy children.

H2: Non-monosymptomatic In postural stabilization in children with enuresis, diaphragmatic breathing is not active compared to healthy children.

H3: Diaphragmatic breathing is not active in postural stabilization in children with daytime Urinary Incontinence compared to healthy children.

One of our aims in this study is to realize the importance of the diaphragm.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with urinary incontinence

  * Being between the ages of 5 -18
  * Accepting participation in the research,

Exclusion Criteria:

* • Less than 5 years old,

  * With spina bifida,
  * Having frequent urinary tract infections,
  * Having a neurological disease,
  * Having a concomitant chronic disease,
  * Cognitive affect,
  * Having mental retardation,
  * Having undergone orthopedic surgery before,
  * In addition to nocturnal incontinence, overactive bladder, delayed voiding, underactive bladder, dysfunctional voiding, bladder outlet obstruction, stress urinary incontinence, vaginal reflux, giggle incontinence, bladder neck dysfunction, neurogenic bladder, urgency
  * Those who do not agree to participate

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study will be conducted with children diagnosed with urinary incontinence in Kırıkale University Medical Faculty Hospital.
Sampling Method: Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2021-02-05 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Scale in Children with Urinary Incontinence (PIN-Q) | through study completion, an average of six months
  It consists of 20 questions. Children are asked to rate each question between 0 and 4 (0=no, 1=never, 2=sometimes, 3=often, 4=always). The total score of the scale ranges from 0 to 80 points. An increase in the total score means that the quality of life of the child is negatively affected.
Voiding Disorders Symptom Score (IBSS) | through study completion, an average of six months
  It measures the severity of children's voiding disorder symptoms. It consists of 14 questions in total. The 13 questions of the questionnaire evaluate symptoms related to daytime incontinence, symptoms related to nocturnal incontinence, frequency of urination in one day, presence of constipation and various urinary incontinence related symptoms. The 14th question evaluates the impact on quality of life in relation to these symptoms.The total score of the scale ranges from 0 to 35 points. An increase in the total score means that the severity of voiding disorders symptom severity increases.
Dynamic Neuromuscular stabilization (DNS) | through study completion, an average of six months
  In the DNS approach, the dual function of the diaphragm, namely respiratory and postural function, is evaluated.
POWERbreathe K5 | through study completion, an average of six months
  It is a respiratory muscle force measurement device. It is designed to match dynamic changes in respiratory muscle strength throughout the breath. S-index (Inspiratory muscle strength), will be evaluated.
POWERbreathe K5 | through study completion, an average of six months
  It is a respiratory muscle force measurement device. It is designed to match dynamic changes in respiratory muscle strength throughout the breath. Maximum inspiratory pressure (MIP) will be evaluated.
POWERbreathe K5 | through study completion, an average of six months
  It is a respiratory muscle force measurement device. It is designed to match dynamic changes in respiratory muscle strength throughout the breath. Volume (Volume (V)) will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Sümeyra KAPUCU, PT, Study Director — Graduate student at Kırıkkale University; Meral SERTEL, Assoc. Prof., Study Chair — Associate professor at Kırıkkale University; Yaşar KANDUR, Assoc. Prof., Principal Investigator — Kırıkkale University, Faculty of Medicine, Pediatric Nephrology Specialist
Locations (1):
- Kirikkale University Faculty of Medicine, Kırıkkale, Turkey (Türkiye)